Protocol: Evaluation of oral condition and the effect of dental treatment on physical

parameters of athletes

Researcher: Caio Vinicius G. Roman Torres

Approval of the Research Ethics Committee in Brazil: 93416718.1.0000.0081

Approval date: 09/August/2018

Informed Consent Form

PROTOCOL: Assessment of oral condition and the effect of dental treatment on physical

parameters of athletes

These clarifications are being presented to request your free and voluntary participation, in the

project Assessment of oral condition and the effect of dental treatment on the physical parameters

of athletes, from the Dentistry Course of the University Santo Amaro - UNISA, which will be

carried out by the researcher Caio Vinicius Gonçalves Roman Torres. The main objective of the

present study will be to evaluate the oral condition and to propose dental treatment according to

the needs for the athletes linked to the Faculty of Physical Education of the University Santo

Amaro. You are being invited to participate in the evaluations and receive instructions on oral

hygiene and, according to the needs presented, you can be referred for treatment at the Dental

Clinic of UNISA. The guests included in the evaluations must follow the following sequence of

evaluations: anamnesis of the participating athletes; clinical examination; assessment of

individual treatment needs; physical exams; instructions for oral hygiene and periodontal

treatment; new clinical and physical exams. No procedure to be performed is experimental, all

are procedures recognized in the literature, which promote improvement in oral conditions.

Periodontal treatment should be performed under local anesthesia, and offers minimal risks or

discomfort for individuals, due to the local anesthesia to be applied and the procedure for root

coronal scraping. In the case of painful symptoms, all individuals will be advised to seek care at

UNISA with Prof. Dr. Caio V. G. Roman Torres at established times during the initial

consultations. We believe that individuals with oral inflammation / infection, the physical

performance should be higher after performing periodontal therapy. Periodontal disease can

influence fatigue and difficulty in recovering from injuries, variables that are so important in an

athlete's life. All participants will have dental follow-up for the treatment of periodontal disease

and when they present other oral problems, they should be referred to the UNISA Dental Clinic

for proper treatment. All participants will receive oral hygiene instructions and explanations about

oral diseases. Access is guaranteed, at any stage of the study, to the professionals responsible for

the research to clarify any doubts or information about the partial results of the research, when in

open studies, or results that are known to the researchers.

The responsible researcher is Prof. Caio Vinicius Gonçalves Roman Torres, which can be found

at Rua Prof. Enéas de Sigueira Neto, 340, Jardim das Imbuías, SP, Telephone (s) 011 2141-8502.

If you have any concerns or doubts about research ethics, please contact the Research Ethics

Committee (CEP-UNISA) - Rua Prof. Enéas de Siqueira Neto, 340, Jardim das Imbuías, SP - Tel

.: 2141-8687.

You are guaranteed your freedom to withdraw consent at any time and stop participating in the

study, without prejudice to the continuity of any benefit you have obtained from the Institution,

before, during or after the period of this study.

The information obtained by the researchers will be analyzed together with that of other

participants, and the identification of none of them will not be disclosed.

There are no personal expenses for the participant at any stage of the study, including exams and

consultations. There is also no financial compensation related to your participation. If there is any

additional expense, it will be absorbed by the research budget.

Pesquisador Responsável: Caio Vinicius Gonçalves Roman Torres - Rua Prof. Enéas de Siqueira Neto, 340, Jardim das Imbuías, SP – Tel.: 13-991304774

In the case of personal injury, directly related to the procedures of this study (proven causal link), at any time, the participant is guaranteed respect for his legal rights, as well as seeking compensation for eventual damages. One copy of this Consent Form will remain in your possession. Sao Paulo, / / Prof. Dr. Caio Vinicius Gonçalves Roman Torres If you agree to participate in this survey, sign in the space specified below and put your name and your identification number. Name: Doc. Identification: ..... I declare (amos) that I obtained (s) appropriately and voluntarily the Free and Informed Consent

of this participant (or of the legal representative of this participant) to participate in this study, as recommended by Resolution CNS 466, of December 12, 2012, IV .3 to 6.

| Signature of the researcher responsible for the study Date // |
|---------------------------------------------------------------|
| Signature of other researchers Date // |